CLINICAL TRIAL: NCT04318158
Title: A Comparative Study of Dexmedetomidine Versus Fentanyl as Adjuvants to Bupivacaine in Ultrasound Guided Transversus Abdominis Plane Block in Patients Undergoing Radical Cystectomy
Brief Title: Dexmedetomidine Versus Fentanyl as Adjuvants to Bupivacaine in Ultrasound Guided Transversus Abdominis Plane Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Dina Mahmoud Fakhry, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Management, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMBSUREC/08032020/Fakhry
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Pain
Keywords: Dexmedetomidine; Fentanyl; Bupivacaine; Transversus Abdominis Plane Block
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Dexmedetomidine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group(B) (Experimental): Patients will receive single shot US guided TAP block using 20 ml bupivacaine 0.25% on each side.
  Interventions: Drug: Bupivacaine
- Group(BD) (Active Comparator): Patients will receive single shot US guided TAP block using 20 ml bupivacaine 0.25% + 50 µg dexmedetomedine on each side.
  Interventions: Drug: Dexmedetomidine
- Group(BF) (Active Comparator): Patients will receive single shot US guided TAP block using 20 ml bupivacaine 0.25% + 50 µg fentanyl on each side.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Bupivacaine — single shot US guided TAP block using 20 ml bupivacaine 0.25%.
  Other Names: Sunnypivacaine
  Arms: Group(B)
Drug: Dexmedetomidine — Single shot US guided TAP block using 20 ml bupivacaine 0.25% + 50 µg dexmedetomedine on each side.
  Other Names: Precedex
  Arms: Group(BD)
Drug: Fentanyl — Single shot US guided TAP block using 20 ml bupivacaine 0.25% + 50 µg fentanyl on each side.
  Other Names: Fentanyl hameln
  Arms: Group(BF)

SUMMARY:
The aim and objective of this study is to compare dexmedetomidine and fentanyl as adjuvants to bupivacaine in ultrasound guided TAP block analgesia in patients undergoing radical cystectomy as regarding postoperative analgesic efficacy.

DETAILED DESCRIPTION:
Radical cystectomy with pelvic lymph node dissection is the gold standard treatment for muscle invasive bladder cancer and is associated with a high risk of complications. Management of the postoperative pain is important to decrease the length of stay in the hospital and the risk of morbidity. Multimodal analgesia management is utilized for pain observed in the postoperative period.As part of a multimodal analgesic regimen, a peripheral nerve block can decrease opioid consumption, providing more effective analgesia with fewer adverse effects.TAP block is a relatively new regional anesthesia technique that provides analgesia to the parietal peritoneum, as well as skin and muscles of the lower anterior abdominal wall. Dexmedetomidine and fentanyl have been used as adjuvants to local anesthetics in different surgeries to provide superior analgesia and to improve the duration of the block.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes.
* ASA grade I and II.
* Age between 50-70 years.
* Elective open radical cystectomy.

Exclusion Criteria:

* Any history or signs of cardiac, hepatic and renal failure.
* Patients with coagulopathy or under anticoagulation therapy.
* Infection near the site of needle insertion.
* Morbid obesity (BMI>40 kg/m2).
* History of allergic reactions to any of the study medications.
* Previous abdominal surgery.
* Patients with any neurological or neuromuscular disorder or history of seizures.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
The time for first rescue analgesia after the TAP block. | first 24 hours after block.
  Postoperative analgesia duration.

SECONDARY OUTCOMES:
the total dose of rescue analgesia after TAP bock. | first 24 hours after block.
  Postoperative analgesia consumption.
VAS for pain. | 0, 2, 4, 6, 12 and 24 hours postoperatively.
  Postoperative pain at rest and movement.

REFERENCES:
- [Derived] Kassim DY, Mahmoud HE, Fakhry DM, Mansour MA. Comparative study of dexmedetomidine versus fentanyl as adjuvants to bupivacaine in ultrasound-guided transversus abdominis plane block in patients undergoing radical cystectomy: a prospective randomised study. BMC Anesthesiol. 2022 Nov 7;22(1):340. doi: 10.1186/s12871-022-01877-1. PMID 36344917